CLINICAL TRIAL: NCT02518698
Title: Treatment Patterns in Castrate Resistant Prostate Cancer Patients With Bone Metastases
Brief Title: Treatment Patterns in Castrate Resistant Prostate Cancer Patients With Bone Metastases in a Medicare Population
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18273
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: Castrated resistant prostate cancer; Patients with bone metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1 / Treatment patterns: Patients with castrated resistant prostate cancer and bone metastases
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Therapies used to treat prostate cancer and more specifically castrate resistant prostate cancer inclusively Xofigo (Radium-223 dichloride, BAY88-8223)

SUMMARY:
The goal of the study is to provide a detailed description of treatments for CRPC (Castrate Resistant Prostate Cancer) patients with bone metastases and the resource utilization and costs associated with that diagnosis and subsequent treatments.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis for bone metastases for members diagnosed with prostate cancer found in the claims data during the identification period
* Members age ≥ 55 to 89 years at index
* Medicare members with medical and pharmacy coverage; and
* Continuously enrolled during the pre- and post-index periods.

Exclusion Criteria:

* Member with diagnosis of any other cancer (excluding melanoma (ICD-9 172.x) and other metastases (ICD-9 198.x)) before the index date; and
* Members age ≥ 89 years of age at index date

Ages: 55 Years to 88 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Castrated resistant prostate cancer patients with bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 1163 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival of mCRPC patients | Up to 24 months
  mCRPC: Metastatic castrate-resistant prostate cancer
Number of skeletal related events (SREs) of the mCRPC patients | Up to 30 months
Type of skeletal related events (SREs) of the mCRPC patients | Up to 30 months
Number of patients with mCRPC with bone metastases | Up to 24 months
Type of treatments associated with mCRPC | Up to 24 months
  Treatments could include chemotherapy or bone radiation
Duration for each treatment identified | Up to 30 months
Distribution of providers by treatment | Up to 30 months
  Distribution of treatments for mCRPC patients will be tracked by the type of provider (oncologist, versus urologist, versus radiation oncologist, etc)
Clinical and demographic characteristics of the mCRPC patients | Up to 12 months
  Gender, age, geographical region and race/ethnicity, Key comorbidities will also be documented using the Deyo-Charlson Comorbidity Index (DCCI); laboratory results for Prostate-Specific Antigen (PSA) and alkaline phosphatase (ALP) testing using laboratory claims; Rx utilization including opioid use
Treatment patterns of mCRPC patients with bone metastases | Up to 30 months
Progression of the disease of mCRPC patients | Up to 12 months

SECONDARY OUTCOMES:
All-cause healthcare resource utilization for mCRPC patients | Up to 30 months
  Using all post-index medical and pharmacy claims, compute the count of physician office visits, outpatient services, inpatient stay, length of inpatient stay, ancillary services, and count of pharmacy claims
mCRPC-specific healthcare resource utilization for mCRPC patients | Up to 30 months
  Healthcare resource utilization will be measured using all post-index medical and pharmacy claims to create counts for physician office visits, outpatient services, inpatient stay, length of inpatient stay, ancillary services and counts of pharmacy claims
All-cause healthcare costs for mCRPC patients | Up to 30 months
  Healthcare costs will be determined using all post-index medical and pharmacy claims. The all-cause total (medical + pharmacy), medical and pharmacy costs will be computed. A family of general linear model analysis will be performed (medical, pharmacy, and total costs)
mCRPC-specific healthcare costs for mCRPC patients | Up to 30 months
  Healthcare costs will be determined using all post-index medical and pharmacy claims where a diagnosis of mCRPC appears in any of the nine diagnosis positions. The mCRPC specific total (Medical + pharmacy), medical and pharmacy costs associated with these claims will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Louisville, Kentucky, United States